CLINICAL TRIAL: NCT02502903
Title: Safety, Tolerability and Activity of BIVV009 in Healthy Volunteers and Patients With Complement-mediated Disorders. A Single/Multiple Ascending Dose Phase 1 Study.
Brief Title: Safety, Tolerability and Activity of BIVV009 in Healthy Volunteers and Patients With Complement Mediated Disorders
Acronym: BIVV009-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Collaborators: Celerion Clinical Research GmbH (Unknown); Assign Data Management and Biostatistics GmbH (Other); ABF Pharmaceutical Services GmbH (Industry); Quest Diagnostics-Nichols Insitute (Industry); Covance (Industry); PPD Laboratories - Virginia (Unknown); Softworld Inc. - Cambridge, MA (Unknown)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTS16214; BIVV009-01 (Other: Bioverativ Therapeutics Inc.); 2014-003881-26 (EudraCT Number)
Record Dates: First submitted 2015-07-07; First posted 2015-07-20 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Bullous Pemphigoid (BP); Cold Agglutinin Disease (CAD); Warm Autoimmune Hemolytic Anemia (WAIHA); End-stage Renal Disease (ESRD)
MeSH Terms: conditions — Pemphigoid, Bullous; Anemia, Hemolytic, Autoimmune; Kidney Failure, Chronic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part A (Placebo Comparator): Single ascending dose (SAD) in NHVs, 7 cohorts, BIVV009 by IV infusion (0.3,1, 3, 10, 30, 60, or 100 mg/kg) or placebo.
  Interventions: Drug: BIV009; Other: Placebo
- Part B (Placebo Comparator): Multiple ascending dose (MAD) in NHVs, 2 cohorts, 4 weekly IV doses of BIVV009 (30 or 60mg/kg) or placebo.
  Interventions: Drug: BIV009; Other: Placebo
- Part C (Experimental): Multiple dose (MD) in a single cohort of patients with various complement-mediated disorders. All patients in Part C will receive a single IV test dose of BIVV009 of 10 mg/kg followed by 4 weekly doses of 60 mg/kg.
  Interventions: Drug: BIV009
- Part E (Experimental): Multiple dose (MD) in a single cohort of patients with cold agglutinin disease previously treated with BIVV009. All patients in Part E will receive a single IV test dose at week 0, week 1, and every 2 weeks thereafter until EOT. Patients who weigh less than 75 kg will receive fixed doses of 6.5 grams of BIVV009; patients who weigh 75 kg or more will receive fixed doses of 7.5 grams of BIVV009. Dose will be increased from 6.5g to 7.5g dose level if patients current weight is >= 75 kg and there is evidence of hematologic breakthrough OR patients current weight is >= 75 kg and there has been at least a 10 percent increase from the patients last recorded weight. Dose will be decreased from 7.5g to 6.5g for patients whose last weight was >= 75 kg and current weight decreased to < 75 kg. Dose decrease will require Sponsor approval.
  Interventions: Drug: BIV009

INTERVENTIONS:
Drug: BIV009
Other: Placebo
  Other Names: saline solution 0.9 %
  Arms: Part A; Part B

SUMMARY:
Prospective, double-blind, randomized, placebo-controlled First-In-Human study with four sub-parts: Part A, a single ascending dose study (SAD) in normal human volunteers (NHVs), Part B, a multiple ascending dose study (MAD) in NHVs, Part C, a multiple dose (MD) study in patients with a complement-mediated disorder, and Part E, a multiple dose (MD) study in patients with cold agglutinin disease previously treated with BIVV009 within the scope of a BIVV009 clinical trial or named patient program use. Note: For parts A-C as well as at the start of part E, study drug was named TNT009. The study drug name is changed to BIVV009 with final version Final 15.0 of the clinical study protocol.

DETAILED DESCRIPTION:
Study TNT009-01 (parts A-C)/ BIVV009 (part E) is a First in Human (FIH) study that uses an Integrated Protocol Design. This Phase 1 study protocol will comprise three sub-parts: a Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) study in normal male and female human volunteers (NHVs), and a Multiple Dose (MD) study in patients with various complement-mediated disorders not confined to a single disease or therapeutic area. Although these patients represent a population with a diverse set of clinical diagnoses they are united by a common mechanism of disease matched to the mechanism of action of BIV009. Several key safety measures have been incorporated into the design of this study, including use of Sentinel Dosing Groups and an independent Data Safety Monitoring Board (DSMB), as well as an appropriate program of prophylactic vaccinations and clinical biomarker surveillance related to the risks potentially associated with inhibition of the complement system. To allow access of BIVV009 to CAD patients where successful treatment effect has been observed and to allow re-initiation of BIVV009 to previously treated CAD patients, Part E has been added to both continued access to study drug in this subset of study patients, and to further characterize the safety and efficacy to BIVV009.

ELIGIBILITY:
Inclusion Criteria:

Part A/B:

* healthy male or female volunteers, age >= 18 years old
* if female, must be post-menopausal, surgically sterilized, or willing/able to use dual, redundant methods of contraception (e.g., barrier plus oral contraceptives) throughout the study
* previously vaccinated against encapsulated bacterial pathogens (Neisseria meningitidis, Haemophilus influenzae, and Streptococcus pneumoniae) or willing to undergo vaccination
* able to comprehend and to give informed consent
* able to co-operate with the investigator, to comply with the requirements of the study, and to complete the full sequence of protocol-related procedures

Part C:

* male or female, age >=18 years old
* if female, must be post-menopausal, surgically sterilized, or willing/able to use dual, redundant methods of contraception (e.g., barrier plus oral contraceptives) throughout the study
* previously vaccinated against encapsulated bacterial pathogens (Neisseria meningitidis, Haemophilus influenzae, and Streptococcus pneumoniae) or willing to undergo vaccination
* able to comprehend and to give informed consent
* able to co-operate with the investigator, to comply with the requirements of the study, and to complete the full sequence of protocol-related procedures
* History of one of the following complement-mediated disorders:

  * bullous pemphigoid (BP)
  * cold agglutinin disease (CAD)
  * warm autoimmune hemolytic anemia (WAIHA)
  * active Antibody-Mediated Rejection (AMR) (acute or chronic) after kidney transplantation
* If CAD, by medical history within the 3 months preceding enrollment, and again at the screening visit:

  - Has hemoglobin < 11.0 g/dL
* If AMR:

  * is >= 180 days post-kidney transplantation with biopsy-proven late AMR
  * has a functioning kidney graft with epidermal growth factor receptor (eGFR) >= 20ml/min/1.73m^2
  * has evidence of late, active AMR (acute or chronic) present on renal allograft biopsy:
  * molecular signature indicating AMR (molecular AMR score > 0.2)
  * morphological and immunohistochemical findings consistent with AMR according to the criteria of the Banff 2013 classification
  * morphological findings consistent with an active rejection process: presence of glomerulitis (g score > 0) and / or peritubular capillaritis (ptc score > 0)
* has immunoglobulin G (IgG) type donor-specific antibody (DSA) present in serum (at time of renal allograft biopsy) with MFI > 1000 in single antigen bead assays
* is willing and able to take routine antibiotic prophylaxis with ciprofloxacin

Part E:

* male or female, age >= 18 years old
* Body weight of >=39 kg at Screening
* history of cold agglutinin disease (CAD) and previously treated with BIVV009 in a BIVV009 clinical trial or named patient program use
* For subjects currently being treated in a BIVV009 named patient program:

  - Evidence of treatment response
* For subjects previously treated in a BIVV009 clinical trial or named patient program not currently receiving BIVV009:

  * Prior evidence of treatment efficacy and hemoglobin <=10.5 g/dL at Screening or Visit 1 (Day 1) or
  * Successful treatment of underlying malignancy or warm autoimmune hemolytic anemia as defined as either:
  * Bone marrow biopsy without evidence of overt hematologic malignancy within the prior 3 months
  * IgG Direct Antiglobulin Test with <=1+ at Screening Visit
  * active hemolysis, with total bilirubin > upper limit of normal (ULN) at the Screening Visit or Visit 1 (Day 1)
* adequate IV access
* negative hepatitis panel (including hepatitis B surface antigen and hepatitis C virus antibody), negative human immunodeficiency virus (HIV) antibody screen and no further clinically significant infection (e.g., pneumonia) at Screening
* if female, must be post-menopausal, surgically sterilised or willing and able to use highly effective methods of birth control throughout the study and for 9 weeks after the last administration of study drug
* able to comprehend and to give informed consent

Exclusion Criteria:

Part A/B:

* clinically significant medical history or ongoing chronic illness that would jeopardize the safety of the subject or compromise the quality of the data derived from his/her participation in this study
* clinically relevant infection of any kind within the preceding month
* clinically relevant abnormal findings on physical examination or clinically relevant laboratory abnormalities
* history of infusion hypersensitivity, allergic or anaphylactic reactions to other therapeutic proteins
* substance abuse, mental illness, or any reason that makes it unlikely in the judgment of the Investigator for the subject to be able to comply fully with study procedures
* use of medication during 2 weeks before the start of the study, which in the judgment of the investigator may adversely affect the subject's welfare or the integrity of the study's results (excluding hormonal contraception in female subjects)
* females who are pregnant (positive pregnancy test at screening or during study phase), lactating, or, if having reproductive potential, are considered potentially unreliable with respect to contraceptive practice
* concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to treatment start
* body weight > 98 kg for all subjects in all dose cohorts other than the 100 mg/kg dose cohort of Part A, for which the body weight upper limit is 58 kg

Part C:

* active acute or chronic viral, bacterial, fungal, or mycobacterial infection, or history of same within preceding month
* autoimmune disorder other than the complement-mediated disorders listed in the Inclusion Criteria
* known malignancy (other than locally limited, previously surgically removed basal cell carcinoma of the skin, lymphoproliferative disorders causally related to the complement-mediated diseases under study, etc.)
* clinically significant hepatobiliary disorder
* history of infusion hypersensitivity, allergic or anaphylactic reactions to other therapeutic proteins
* substance abuse, mental illness, or any reason that makes it unlikely in the judgment of the Investigator for the subject to be able to comply fully with study procedures
* females who are pregnant (positive pregnancy test at screening or during study phase), lactating, or, if having reproductive potential, are considered potentially unreliable with respect to contraceptive practice
* concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to treatment start
* body weight >98 kg
* Solely for kidney transplantation patients with AMR:

  * acute graft dysfunction within preceding 1 month
  * rejection treatment within preceding 1 month
  * morphological or molecular features of T cell-mediated rejection on renal allograft biopsy
  * contraindication to ciprofloxacin

Part E:

* concurrent or prior treatment within the 3 months immediately preceding the Screening Visit (although more remote prior treatment is permitted) with rituximab, azathioprine, or other immune-suppressive therapy (concurrent treatment with corticosteroids is allowed if on stable dose <= 10mg/day prednisone for previous 3 months)
* concurrent or prior treatment within the 6 months immediately preceding the Screening Visit with rituximab combination therapy or other cytotoxic therapy (e.g., fludarabine, bendamustine, cyclophosphamide, ibrutinib or any other cytotoxic drugs)
* For subjects previously treated in a BIVV009 clinical trial not currently receiving BIVV009:

  * Ferritin below the lower limit of normal. Concurrent treatment with iron supplementation is permitted if the patient has been on a stable dose for the previous 4 weeks
  * Erythropoietin deficiency. Concurrent treatment with erythropoietin is permitted if the patient has been on a stable dose for the previous 6 weeks
  * Clinical diagnosis of systemic lupus erythematosus (SLE); or other autoimmune disorders with anti-nuclear antibodies at Screening
* Clinically significant medical history or ongoing illness that is new or progressed since last BIVV009 therapy that would jeopardize the safety of the patient or compromise the quality of the data derived from his/her participation in this study (as determined by the Investigator [or designee] at Screening.
* concurrent plasma exchange therapy
* females who are pregnant (positive pregnancy test at screening or during study phase), lactating, or, if having reproductive potential, are considered potentially unreliable with respect to contraceptive practice
* concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to treatment start or during the entire study
* history of infusion hypersensitivity, or allergic or anaphylactic reactions to BIVV009.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Drug-related Adverse Event profile of BIVV009 | 6 weeks
  Serious and Non-Serious adverse events probably or possibly attributable to BIVV009

SECONDARY OUTCOMES:
Pharmacokinetic profile of BIVV009 | 6 weeks
  Tmax, Cmax, Area under curve (AUC) and T1/2
Classical pathway complement system activity | 6 weeks
  inhibition by BIVV009 of the complement system classical pathway measured by the WIESLAB® assay
Complement System-Related biomarkers | 6 weeks
  e.g. CH50
Coagulation System-Related biomarkers | 6 weeks
  e.g. Fibrin D-dimer
Disease-Related Biomarkers | 6 weeks
  e.g. Haptoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Vo A, Ammerman N, Jordan SC. New Therapies for Highly Sensitized Patients on the Waiting List. Kidney360. 2024 Aug 1;5(8):1207-1225. doi: 10.34067/KID.0000000000000509. Epub 2024 Jul 12. PMID 38995690
- [Derived] Jager U, D'Sa S, Schorgenhofer C, Bartko J, Derhaschnig U, Sillaber C, Jilma-Stohlawetz P, Fillitz M, Schenk T, Patou G, Panicker S, Parry GC, Gilbert JC, Jilma B. Inhibition of complement C1s improves severe hemolytic anemia in cold agglutinin disease: a first-in-human trial. Blood. 2019 Feb 28;133(9):893-901. doi: 10.1182/blood-2018-06-856930. Epub 2018 Dec 17. PMID 30559259
- [Derived] Eskandary F, Jilma B, Muhlbacher J, Wahrmann M, Regele H, Kozakowski N, Firbas C, Panicker S, Parry GC, Gilbert JC, Halloran PF, Bohmig GA. Anti-C1s monoclonal antibody BIVV009 in late antibody-mediated kidney allograft rejection-results from a first-in-patient phase 1 trial. Am J Transplant. 2018 Apr;18(4):916-926. doi: 10.1111/ajt.14528. Epub 2017 Oct 31. PMID 28980446
- [Derived] Muhlbacher J, Jilma B, Wahrmann M, Bartko J, Eskandary F, Schorgenhofer C, Schwameis M, Parry GC, Gilbert JC, Panicker S, Bohmig GA. Blockade of HLA Antibody-Triggered Classical Complement Activation in Sera From Subjects Dosed With the Anti-C1s Monoclonal Antibody TNT009-Results from a Randomized First-in-Human Phase 1 Trial. Transplantation. 2017 Oct;101(10):2410-2418. doi: 10.1097/TP.0000000000001804. PMID 28926521
- [Derived] Derhaschnig U, Gilbert J, Jager U, Bohmig G, Stingl G, Jilma B. Combined integrated protocol/basket trial design for a first-in-human trial. Orphanet J Rare Dis. 2016 Oct 4;11(1):134. doi: 10.1186/s13023-016-0494-z. PMID 27716293